CLINICAL TRIAL: NCT06007560
Title: Aerobe Cycling Training in Women With Unexplained Recurrent Pregnancy Loss
Acronym: HMOVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Tess Meuleman, Principal Investigator, Radboud University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HMOVE
Record Dates: First submitted 2022-11-29; First posted 2023-08-23 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Pregnancy Loss
Keywords: Natural Killer cells
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- <80% eNK (Other): Women with low eNK bright cell numbers, defined as <80% of the total endometrial NK cell population
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Aerobe cycling training consisting of 12-weeks of HR-controlled training at 50-60% of VO2max (maximal oxygen uptake) for 1 hour, for 2 times (week: 1-6) to 3 times (week: 7-12) per week

SUMMARY:
In 50% of women with recurrent pregnancy loss (RPL) miscarriages are unexplained, therefore no therapeutic intervention is possible. In a pilot study, women with unexplained RPL showed less endometrial NK cells (eNK) compared to women with a previously uncomplicated pregnancy. It is known that eNK cells are important for embryo implantation during early pregnancy. Investigators presume that high sympathetic activity in these women is related to eNK cell number, function and phenotype and that exercise is an effective intervention to lower sympathetic activity and to influence the immune system, as especially peripheral NK cells have been assumed to be responsive to physical training. The investigators hypothesize that moderate exercise can lower the adrenergic tone of the sympathetic nervous system hereby influencing endometrial NK cells in women with RPL and eventually pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

* RPL defined as 2 or more unexplained pregnancy losses from the time of conception until 24 weeks of gestation, known cause for the miscarriages are the presence of thyroid abnormalities, anti-phospholipid syndrome, uterine malformation, and abnormal parental karyotype according to international guideline.
* Couples should not be aiming to conceive during the time course of the exercise intervention.

Exclusion Criteria:

* Age above 40 years
* BMI above 40
* Current use of immunosuppressive or biological drugs
* Current use of hormone conceptive
* HIV positivity
* Current or recent (<2 weeks) symptomatic genital infection such as chlamydia, gonorroa, or pelvic inflammatory disease
* Pre-existent diabetes mellitus, autoimmune disease or overt cardiovascular disease
* Vaccination (i.e Covid) within 1 month prior to or during sampling and intervention
* New pregnancy at time of measurements, breastfeeding
* Current or recent (<2-3 months ago) pregnancy
* (Physical) inabilities to follow moderate aerobe cycling training
* Participants who are not capable of signing the informed consent

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
CD56 endometrial NK cell frequency | 3 months
  Change in CD56 eNK cell frequency measured as percentage of total lymphocyte or total CD56 population by flowcytometry.
CD56 endometrial NK cell function | 3 months
  Change in CD56 eNK cell function measured as percentage of CD56 degranulation by flowcytometry.

SECONDARY OUTCOMES:
CD56 endometrial NK cell phenotype | 3 months
  Change in CD56 eNK cell phenotype measured as percentage of (sub)population or mean fluorescent intensity respectively by flowcytometry.
CD56 peripheral NK cell frequency | 3 months
  Change in CD56 pNK cell frequency measured as percentage of total lymphocyte or CD56 population by flowcytometry.
CD56 peripheral NK cell function | 3 months
  Change in CD56 pNK cell function measured as percentage of CD56 degranulation by flowcytometry.
CD56 peripheral NK cell phenotype | 3 months
  Change in CD56 pNK cell phenotype measured as percentage of (sub)population or mean fluorescent intensity respectively by flowcytometry.
Vaginal microbiome | 3 months
  Change in taxonomic classification of vaginal microbiota of different subtypes but also classified in clustering of different subtypes.
Metabolic syndrome parameters I | 3 months
  Change in cm waist circumference.
Metabolic syndrome parameters II | 3 months
  Chance in mmHg blood pressure, both systolic as diastolic.
Metabolic syndrome parameters III | 3 months
  Change in concentration (mg/dL) triglyceride.
Metabolic syndrome parameters IV | 3 months
  Change in concentration (mg/dL) cholesterol levels.
Metabolic syndrome parameters V | 3 months
  Change in concentration (mg/dL) blood sugar levels.
Sympathetic activity | 3 months
  Change in baroreceptor sensitivity in ms/mmHg.
Uterine blood flow | 3 months
  Change in pulsatility index, lower indicates better outcome.
Physical fitness | 3 months
  Change in VO2max.
Pregnancy rate and live birth rate after one year of intervention, higher rater indicate better outcome. | 3 months
  Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Tess Meuleman, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Maastricht UMC+, Maastricht
  - Radboud UMC, Nijmegen

IPD SHARING:
Plan to Share IPD: No
On reasonable special request only.